CLINICAL TRIAL: NCT00405626
Title: Phase 2 Study of the Effect of Bellis Perenis and Arnica Montana on Post Partum Hemmorhage
Brief Title: Double Blind Placebo Controlled Bellis Perenis and Arnica Montana as a Drug for PPH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hompostpartum-HMO-CTIL
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-02

CONDITIONS: Hemorrhage
Keywords: post partum hemmorhage,Arnica montana,Bellis Perenis
MeSH Terms: conditions — Hemorrhage

INTERVENTIONS:
Drug: Bellis Perenis ,Arnica montana

SUMMARY:
To look at the antihemmorhagic effect of 2 homeopathic drugs in women post delivery Bellis Perenis and Arnica montana

DETAILED DESCRIPTION:
To look at the antihemmorhagic effect of 2 homeopathic drugs in women post delivery Bellis Perenis and Arnica montana compare it with placebo

ELIGIBILITY:
Inclusion Criteria:

* healthy women during delivery

Exclusion Criteria:

* Scarred uterus, multifetal ,multiparty,bleeding problems,cesarean sectons,chorioamnionitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2007-04; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
hemoglobin levels 2 days post partum

SECONDARY OUTCOMES:
pain

CONTACTS AND LOCATIONS:
Overall Officials: David Mankuta, Study Chair — Hadassah University Medical Organization
Locations (1):
- Haddasah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Oberbaum M, Galoyan N, Lerner-Geva L, Singer SR, Grisaru S, Shashar D, Samueloff A. The effect of the homeopathic remedies Arnica montana and Bellis perennis on mild postpartum bleeding--a randomized, double-blind, placebo-controlled study--preliminary results. Complement Ther Med. 2005 Jun;13(2):87-90. doi: 10.1016/j.ctim.2005.03.006. PMID 16036165